CLINICAL TRIAL: NCT04319926
Title: An Open Label, Randomized, Two-treatment, Two-period, Single-dose Study Evaluating the Product Adhesion in Healthy, Adult Subjects Using ZTlido 1.8% Topical System and a Generic Lidocaine Patch 5%.
Brief Title: Adhesion Performance Study of Lidocaine Topical System 1.8% Compared to Generic Lidocaine Patch 5% in Healthy, Adult, Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Scilex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SCI-LIDO-ADH-003
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Healthy
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lidocaine Patch (Sequence T1T2) (Experimental): Subjects receive both lidocaine topical system 1.8% and the generic lidocaine patch 5%. The sequence in which they receive the lidocaine products is determined by random assignment. For subjects in Arm 1, lidocaine 1.8% topical systems are applied in Period 1, and the generic lidocaine 5% patches are applied in Period 2.
  Interventions: Drug: lidocaine topical system 1.8%; Drug: lidocaine patch 5%
- Lidocaine Patch (Sequence T2T1) (Experimental): Subjects receive both lidocaine topical system 1.8% and the generic lidocaine patch 5%. The sequence in which they receive the lidocaine products is determined by random assignment. For subjects in Arm 2, generic lidocaine 5% patches are applied in Period 1, and the lidocaine 1.8% topical systems are applied in Period 2.
  Interventions: Drug: lidocaine topical system 1.8%; Drug: lidocaine patch 5%

INTERVENTIONS:
Drug: lidocaine topical system 1.8% — One topical system is applied to the subject's back for 12 hours.
  Other Names: lidocaine patch 1.8%; ZTlido
Drug: lidocaine patch 5% — One generic lidocaine patch is applied to the subject's back for 12 hours.

SUMMARY:
An open label, randomized, two-treatment, two-period, single-dose study evaluating the product adhesion in healthy, adult subjects using ZTlido 1.8% Topical System and a generic Lidocaine Patch 5%

ELIGIBILITY:
Key Inclusion Criteria:

* Must be healthy based on by medical history, laboratory work, ECG, and physical exam with BMI range between 18.00 and 30.00 kg/m2 inclusive.
* Be at least 18 years of age
* If childbearing potential, use of acceptable form of birth control
* In the case of females of childbearing potential, have a negative serum pregnancy test

Key Exclusion Criteria:

* Allergy or known hypersensitivity to lidocaine, amide-type local anesthetics, or any component of the product formulation
* Any major medical illness 3 months prior or any significant history or ongoing chronic medical illness
* Subjects with conditions that might affect application of the product or its adhesive properties (including psoriasis, eczema, atopic dermatitis, damaged or irritated epidermal layer, and excessive hair or oil on the skin)
* History of addiction, abuse, and misuse of any drug
* Use of local anesthetics of antiarrhythmic drugs (such as tocainide or mexiletine) within 14 days prior to product application

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-07 (Actual); Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
Mean Percent Adhesion | 12 hours post-dose
  Percent adhesion is assessed by laying a transparent sheet the exact size of the product over the top of the product and outlining areas of adhesion with a marker on the transparent sheet. The area excluded from the adhered area will be assessed to determine the degree of lift-off. Adhesion is assessed every 3 hours after product application. Mean percent adhesion is calculated as the sum of scores at each assessment time point divided by the total number of observations.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Luger, MD, Principal Investigator — AXIS Clinicals
Locations (1):
- AXIS Clinicals, Dilworth, Minnesota, United States

REFERENCES:
- [Derived] Gudin J, Webster LR, Greuber E, Vought K, Patel K, Kuritzky L. Open-Label Adhesion Performance Studies of a New Lidocaine Topical System 1.8% versus Lidocaine Patches 5% and Lidocaine Medicated Plaster 5% in Healthy Subjects. J Pain Res. 2021 Feb 23;14:513-526. doi: 10.2147/JPR.S287153. eCollection 2021. PMID 33654425